CLINICAL TRIAL: NCT07053891
Title: LUPKYNIS Drug-use Results Survey
Status: Recruiting | Type: Observational
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 348-101-00044
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — voclosporin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Voclosporin (LUPKYNIS) — In general, for adults, voclosporin should be administered orally at a dose of 23.7 mg BID. The dosage may be appropriately reduced depending on the patient's condition. In principle, at the start of treatment with voclosporin, it should be used in combination with corticosteroids and mycophenolate mofetil.

SUMMARY:
The purpose of this study is to survey the safety of LUPKYNIS in patients with lupus nephritis under actual use conditions. In addition, information on efficacy will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are newly starting administration of LUPKYNIS for lupus nephritis

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in Japan who are planned to be newly started on LUPKYNIS for lupus nephritis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2031-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety Information (Number of Adverse Event) | 3 years from the initiation of LUPKYNIS treatment
  Any untoward medicinal occurrence in a patient or clinical study subject administered a Medicinal Product and which does not necessarily have a causal relationship with this treatment (ICH-E2A Guideline). An Adverse Event can therefore be any unfavorable and unintended sign (e.g. abnormal laboratory finding), symptom, or disease temporally associated with the use of a Medicinal Product (LUPKYNIS), whether or not it is considered causally related to the Medicinal Product.
Safety Information (Types of Special Situations and the Number of Corresponding Cases) | 3 years from the initiation of LUPKYNIS treatment
  Situations related to the use of an Otsuka product which may or may not be associated with an adverse event:
  * Maternal (pregnancy and breastfeeding) or paternal (via semen) exposure;
  * Exposure during breastfeeding;
  * Overdose/Incorrect dosage, misuse, abuse (e.g. patient sharing products); -Medication errors (e.g. patient took wrong dose);
  * Lack of therapeutic efficacy (e.g. the product doesn't work);
  * Occupational exposure (e.g.: nurse administering the product is exposed);
  * Cases of suspected transmission of infectious agents;
  * Use of suspected or confirmed falsified product(s) or quality defect of the product(s);
  * Withdrawal reactions; -Accidental exposure (e.g.: child takes parent's product);
  * Drug-drug/drug-food interactions;
  * Unintentional use of product in a non-approved population (e.g.: pediatric or geriatric population);
  * Disease progression/exacerbation of existing disease.
Safety Information (Number of off-Label Use) | 3 years from the initiation of LUPKYNIS treatment
  Collecting any type of off-Label Use that refers to situations where a product is intentionally used for a medical purpose not in accordance with the authorized product information. Off-label use also includes the intentional use in non-authorized population categories not indicated in the label.
Safety Information (Number of Serious Adverse Event) | 3 years from the initiation of LUPKYNIS treatment
  Any adverse drug experience/event occurring at any dose which
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or prolonged of existing hospitalization
  * results in persistent or significant disability or incapacity
  * is a congenital anomaly/birth defect
  * is medically significant.
Safety Information (Number of Non-serious Adverse Events) | 3 years from the initiation of LUPKYNIS treatment
  All Adverse Events that do not meet the definition of a serious Adverse Event are considered non-serious Adverse Events.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacovigilance Department, Osaka, Osaka, Japan